CLINICAL TRIAL: NCT04929184
Title: Speech Processing in Stuttering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Emily O'Dell Garnett, Research Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00194953; 1R21DC019429-01 (NIH)
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Stuttering; Stuttering, Childhood; Stuttering, Adult
Keywords: Healthy children; Healthy Adults
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adults who stutter (AWS) (Experimental): Participants will have 2 visits.
  Interventions: Behavioral: Speech and non-speech tasks
- Healthy Adults (Other): Participants will have 2 visits.
  Interventions: Behavioral: Speech and non-speech tasks
- Children who Stutter (Experimental): Participants will have 1 visit.
  Interventions: Behavioral: Speech and non-speech tasks
- Healthy Children (Other): Participants will have 1 visit.
  Interventions: Behavioral: Speech and non-speech tasks

INTERVENTIONS:
Behavioral: Speech and non-speech tasks — Participants will complete speech tasks such as listening to and/or producing speech and non-speech sounds.

SUMMARY:
This research is being done to better understand stuttering, specifically how people who stutter may process and/or produce speech. Eligible participants enrolled will complete a variety of computer and speech-based tasks on up to 2 visits.

DETAILED DESCRIPTION:
The study team will update the record to include the secondary identification number once the NIH has released the funds.

ELIGIBILITY:
Inclusion Criteria (adults who do not stutter):

* 18-65 years old
* English as primary language
* Normal speech, language, hearing, cognition

Exclusion criteria: (adults who do not stutter)

* Personal or family history of stuttering
* Major medical or psychiatric illness

Inclusion criteria: (adults who stutter)

* Aged 18-65 years
* English as primary language
* Normal speech, language, hearing, cognition (other than stuttering)
* Currently stutters

Exclusion criteria: (adults who stutter)

* Speech therapy within the past year
* Major medical or psychiatric illness

Inclusion criteria: (children who do not stutter)

* Aged 6 to 17 years
* English as primary language
* Normal speech, language, hearing, cognition

Exclusion criteria: (children who do not stutter)

* Personal or family history of stuttering
* Major medical or psychiatric illness
* Language/motor delay

Inclusion criteria: (children who stutter)

* Aged 6 to 17 years
* English as primary language
* Normal speech, language, hearing, cognition (other than stuttering)
* Currently stutters

Exclusion criteria: (children who stutter)

* Major medical or psychiatric illness
* Language/motor delay

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Phase locking value (PLV) - Session 1 speech tasks | Session 1 (up to 4 hours)
  The degree of synchronization will be measured by computing the PLV between subject's produced speech and the heard speech. The PLV is a vector with a value between 0 and 1 that reflects the phase difference between two signals.
Phase locking value (PLV) - Session 2 speech tasks | Session 2 (up to 4 hours)
  The degree of synchronization will be measured by computing the PLV between subject's produced speech and the heard speech. The PLV is a vector with a value between 0 and 1 that reflects the phase difference between two signals. Session 2 is for adults only.

SECONDARY OUTCOMES:
Phase locking value (PLV) - Non-speech tasks | Session 1 (up to 4 hours)
  The degree of synchronization will be measured by computing the PLV between subject's produced response and the auditorily presented stimuli. The PLV is a vector with a value between 0 and 1 that reflects the phase difference between two signals.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Garnett, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan

IPD SHARING:
Plan to Share IPD: No